CLINICAL TRIAL: NCT04920903
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, First-in-Human, Single- and Multiple-Ascending Dose Study Evaluating the Safety, Tolerability, and Pharmacokinetics of Oral COR588 in Healthy Adult Subjects
Brief Title: A Single and Multiple Ascending Dose Study of COR588
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cortexyme Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: COR588
Record Dates: First submitted 2021-06-04; First posted 2021-06-10 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- COR588 (Experimental)
  Interventions: Drug: COR588
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: COR588 — Increasing doses of COR588 will be administered for cohorts 1-4 in the single ascending dose phase and for cohorts 1-4 in the multiple ascending dose phase.
  Arms: COR588
Drug: Placebo — Placebo will be administered for cohorts 1-4 in the single ascending dose phase and for cohorts 1-4 in the multiple ascending dose phase.
  Arms: Placebo

SUMMARY:
The study is a randomized, double-blind, placebo-controlled, single and multiple ascending dose study to assess the safety and tolerability of COR588 HCl in healthy male and female subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects between 18 to 55 years of age, inclusive (at the time of consent) for Part A;
* Body mass index between 18 and 32 kg/m2, inclusive, at screening and Day -1;
* Participants with no clinically significant abnormal screening results in the opinion of the investigator;
* All screening laboratory parameters (chemistry, hematology, coagulation, urinalysis) within normal limits or considered not clinically significant in the opinion of the investigator. If necessary, in the investigator's opinion, screening labs may be repeated once to confirm the results if error is suspected.
* Women of childbearing potential (WOCBP) must have a negative blood or urine pregnancy test within 24 hours prior to the start of investigational product and must not be breastfeeding, lactating or planning pregnancy during the study period. WOCBP must agree to use an acceptable form of contraception during the treatment period and for at least 30 days after the last dose of investigational product.
* A male subject with a female partner of childbearing potential is eligible to participate if he agrees to use acceptable contraception during the treatment period and for at least 90 days after the last dose of study treatment and refrains from donating sperm during this period;
* Agree to comply with study-specified diet and consume the high-fat breakfast in its entirety (food effect cohort) while confined in the study site;
* Provide signed informed consent prior to any study procedures commencing, understand and comply with the requirements of the study, and be able to communicate with the investigator.

Exclusion Criteria:

* Presence of significant neurological, cardiovascular, hematological, psychiatric, hepatic, gastrointestinal, pulmonary, endocrine, immunologic or renal disease;
* History or presence of malignancy within the past 2 years prior to Day -1 with the exception of adequately treated basal cell or squamous cell carcinoma of the skin;
* History of conditions (e.g., chronic diarrhea or prior abdominal surgery) known to interfere with the absorption, distribution, metabolism, or excretion of drugs;
* Clinically significant acute illness or infection within 14 days prior to Day -1;
* Any surgical procedure within 3 months prior to Day -1, that may interfere with the performance in the study in the judgment of the investigator;
* History or presence of cardiac abnormalities or congenital long QT syndrome;
* Subjects with a QTcF interval >450 msec for males and >470 msec for females at screening or Day -1;
* Any dietary restriction, intolerance, or food allergy that would prohibit the consumption of a high fat breakfast (food effect cohort only);

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2021-08-26 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment emergent adverse events. | Through Day 8 for the single ascending dose phase and through Day 19 for the multiple ascending dose phase.
  Assessment of the incidence and severity of treatment-emergent adverse events.
Changes in chemistry lab measures (Sodium [Na], Blood Urea Nitrogen [BUN], Calcium [Ca], Total bilirubin). | Through Day 8 for the single ascending dose phase and through Day 19 for the multiple ascending dose phase.
  Assessment of changes in serum chemistry measures.
Changes in hematology lab measures (red blood cell count [RBC], hemoglobin [Hgb], hematocrit [Hct]). | Through Day 8 for the single ascending dose phase and through Day 19 for the multiple ascending dose phase.
  Assessment of changes in hematology measures.
Changes in urinalysis lab parameters (pH, specific gravity, glucose). | Through Day 8 for the single ascending dose phase and through Day 19 for the multiple ascending dose phase.
  Assessment of changes in urinalysis parameters.

SECONDARY OUTCOMES:
AUC | To Day 3 for the single ascending dose phase and to Day 11 for the multiple ascending dose phase.
  Area under the concentration-time curve
Cmax | To Day 3 for the single ascending dose phase and to Day 11 for the multiple ascending dose phase.
  Maximum observed drug concentration during a dosing interval
Tmax | To Day 3 for the single ascending dose phase and to Day 11 for the multiple ascending dose phase.
  Time to Cmax

CONTACTS AND LOCATIONS:
Locations (1):
- Nucleus Network Pty Ltd, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No